CLINICAL TRIAL: NCT01584882
Title: Computer-Assisted Guidance for Tobacco Dependence Interventions in Dental Offices
Brief Title: Computer-Assisted Tobacco Interventions in Dental Offices
Acronym: CATI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-062
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2014-07

CONDITIONS: Smoking
Keywords: Clinical decision support (CDS); Tobacco; Behavioral; Dental hygienist; Dentist; Smoking; Electronic health record
MeSH Terms: conditions — Smoking; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Usual care) (No Intervention): Return patients seen within the data collection window in HealthPartners Dental Clinics (new patient exams were excluded) who were documented as using tobacco, specifically cigarettes, at their last dental encounter. Randomization was at the clinic level.
- Tobacco Cessation Tool (CATI Tool) (Experimental): Using Screening for drug use, Brief Intervention, Referral to Treatment (SBIRT) as a model, a 'CATI'[Computer Assisted Tobacco Intervention] tool was designed for the Electronic Dental Record which required assessment of 4 variables for patients reporting cigarettes use: 1) number of cigarettes daily, 2) how soon upon waking the first cigarette was smoked, 3) interest in quitting, and 4) previous quit attempts. Level of dependency was calculated and displayed in the health history using the Heavy Smoking Index. Pop-up provider scripts were generated using rule-based algorithms. Links to printable patient education materials on the quit line and on medications to help quit smoking were embedded in the scripts window. The tool automatically recorded tobacco-cessation details.
  Interventions: Behavioral: CATI Tool

INTERVENTIONS:
Behavioral: CATI Tool — Using Screening for drug use, Brief Intervention, Referral to Treatment (SBIRT) as a model, a CATI tool was designed for the Electronic Dental Record which required assessment of 4 variables for patients reporting cigarettes use: 1) number of cigarettes daily, 2) how soon upon waking the first cigarette was smoked, 3) interest in quitting, and 4) previous quit attempts. Level of dependency was calculated and displayed in the health history using the Heavy Smoking Index. Pop-up provider scripts were generated using rule-based algorithms. Links to printable patient education materials on the quit line and on medications to help quit smoking were embedded in the scripts window. The tool automatically recorded tobacco-cessation details.
  Arms: Tobacco Cessation Tool (CATI Tool)

SUMMARY:
Electronic dental records (EDR) are a potentially powerful tool to incorporate current scientific evidence into clinical practice by providing key information at the point of patient care. The investigators know that disseminating evidence-based guidelines is not sufficient to change clinical practice so innovative approaches need to be tested in dentistry. The composite expertise of the investigators and consultants on this project and a large group practice with multiple clinics utilizing one EDR are essential to address the aims of this study. This project will examine whether dentists and hygienists will assess interest in quitting and deliver a tobacco intervention more frequently when provided with computer assisted guidance compared to a control group. Specifically the investigators will measure the delivery of questions assessing willingness to change and appropriate interventions based on willingness to change by measuring the recording of these activities in the EDR and patient receipt of these recommendations through a phone survey. In addition, the study will do a qualitative assessment of the patient perceived value of the provider-patient encounter to further inform us about patient perception of this interaction. The investigators want to know if dental providers will utilize these tools during the dental encounter. If they are used, the investigators would propose further studies examining smoking cessation rates. The investigators were not able to measure cessation rates due to the short two year timeline of this funding mechanism. This tool has potential application for other clinical topics, which makes this approach very innovative when considering the translation of evidence into the unique clinical practice of dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Adult dental patient presenting for an exam visit whose most recent history reports the patient is a smoker. Patients had to agree to the phone survey.

Exclusion Criteria:

* Research opt out list
* Patients who discontinued the survey prior to completion(considered withdrawals)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Patient report | Within 3 days of the dental encounter
  Patient report of dental providers delivery of:
  1. Screening for tobacco
  2. Discussion of specific strategies to assist the patient with quitting smoking
  3. Referral to a Quitline (toll free number for comprehensive tobacco cessation support)

CONTACTS AND LOCATIONS:
Overall Officials: D. Brad Rindal, DDS, Principal Investigator — HealthPartners Researc Foundation
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- [Derived] Rindal DB, Rush WA, Schleyer TK, Kirshner M, Boyle RG, Thoele MJ, Asche SE, Thyvalikakath T, Spallek H, Durand EC, Enstad CJ, Huntley CL. Computer-assisted guidance for dental office tobacco-cessation counseling: a randomized controlled trial. Am J Prev Med. 2013 Mar;44(3):260-4. doi: 10.1016/j.amepre.2012.10.023. PMID 23415123
- See also: HealthPartners Research Foundation — http://www.hprf.org